CLINICAL TRIAL: NCT00603148
Title: The Role of Platelet Surface α2β1 Integrin Expression as a Risk Factor in Thrombotic and/or Bleeding Complications in Patients Undergoing Invasive Procedures in the Hybrid Cardiac Catheterization/Cardiac Surgery Suite
Brief Title: The Role of Platelet Surface α2β1 Integrin Expression as a Risk Factor in Thrombotic and/or Bleeding Complications
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samuel A. Santoro, Professor and Chair, Pathology, Microbiology & Immunology, Vanderbilt University
Other Study IDs: 060433
Record Dates: First submitted 2007-10-17; First posted 2008-01-28 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Genetic Polymorphism
Keywords: Genetic Polymorphism; Integrin alpha2beta1; Phenotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will begin to define these critical determinants for patients undergoing procedures in the hybrid interventional cardiology/cardiac surgery suite. In future studies, the data obtained from this study will be used to prospectively stratify patients in terms of bleeding verses thrombotic risk to design studies to optimize anticoagulation and anti-platelet therapies in the hybrid setting.

DETAILED DESCRIPTION:
The aim of this study is to test the association of DNA polymorphisms linked to the level of αβ1 integrin expression on platelets with clinical outcome in terms of bleeding or thrombotic complications. The association of polymorphisms in other genes such as GPVI, PAR-1, and COX-2, as well as PLA ½ status, will also be examined and considered in the context of other factors such as medications including IIb/IIIa inhibitors, anticoagulants, type of procedure, obesity smoking status, etc.

Lower levels of platelet surface expression of the α2β1 integrin are associated with an increased risk of bleeding complications following hybrid procedures, especially when the low level of integrin expression is associated with other risk factors that may exacerbate bleeding such as vigorous anti-coagulation, aggressive anti-platelet therapy and other genetic risk factors that contribute to a hemorrhagic phenotype. Conversely, higher level expression of the α2β1 integrin is likely associated with a greater tendency to thrombotic complication that is again modified by other coexisting risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited to the study who are to undergo elective hybrid procedures [percutaneous coronary intervention (PCI) followed by minimally invasive coronary artery bypass graft (CABG) surgery or valve surgery].
* Both male and females will be enrolled in this study.
* The age of the population is 18-70 years old.
* No one ethnic group or gender will be targeted or excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing procedures in a hybrid interventional cardiology/cardiac surgery suite
Sampling Method: Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
genetic determination of bleeding verses thrombotic risk factors in patients undergoing cardiovascular procedures

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A. Santoro, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States